CLINICAL TRIAL: NCT01096693
Title: Effects of Urocortins on Forearm Arterial Blood Flow in Healthy Volunteers
Brief Title: Effects of Urocortins on Forearm Arterial Blood Flow in Healthy Volunteers (Protocol 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SV.Procotol 2
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Vascular Disease; Heart Disease
Keywords: Urocortin 2; Urocortin 3; Astressin 2B; forearm blood flow; plethysmography; vascular; heart failure
MeSH Terms: conditions — Vascular Diseases; Heart Diseases; Heart Failure | interventions — Urocortins; Substance P

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Placebo (Placebo Comparator): In this arm, the response in forearm blood flow to incremental doses of Urocortins 2, 3 and Substance P will be studied co infused with saline placebo.
  Interventions: Drug: Saline placebo
- Response to Urocortin infusion in presence of Astressin 2B (Active Comparator): This arm studies the response to intra arterial infusion of incremental doses of Urocortins 2, 3 and Substance P in the presence or absence of a selective antagonist - Astressin 2B.
  Interventions: Drug: Urocortin 2, Urocortin 3

INTERVENTIONS:
Drug: Urocortin 2, Urocortin 3 — After a 20 minute infusion of intra arterial saline, healthy volunteers will receive ascending doses of intra arterial Urocortin 2 (3.4, 34 and 340 pmol/min to achieve estimated end-organ concentrations of 0.06, 0.6 and 6 µg/L, respectively), Urocortin 3 (3.4, 34 and 340 pmol/min to achieve estimated end-organ concentrations of 0.06, 0.6 and 6 µg/L, respectively) and Substance P (a control endothelium-dependent vasodilator that evokes endogenous t-PA release [2, 4 and 8 pmol/min]). This will be co-infused with either Astressin 2B (in one of the two doses determined from Protocol 1) or saline placebo.
  Bilateral venous blood sampling will be performed at baseline, immediately before the start and after each dose of Urocortin 2 and 3, to later estimate net release of tPA and PAI-1 and for plasma measurements of Urocortins 2 and 3.
  Other Names: Forearm vascular study - Forearm blood flow will be measured using venous occlusion plethysmography at baseline and with each dose of Ucn 2, 3 and Substance P.
  Arms: Response to Urocortin infusion in presence of Astressin 2B
Drug: Saline placebo — After 20 minutes of intra arterial saline infusion, incremental doses of Urocortin 2, 3 and Substance P will be administered (in doses similar to Active comparator arm), co infused with saline placebo.
  Bilateral venous blood samples will be taken at baseline, immediately before the start of Ucn2/Ucn3 infusion and at the end of each dose of Ucn2/Ucn3 for subsequent calculation of net release of t-PA and PAI-1.
  Other Names: Forearm vascular study - Bilateral forearm blood flow will be measured at baseline and after each dose of Ucn 2, 3 and Substance P.
  Arms: Saline Placebo

SUMMARY:
Impairment of the heart's pumping capacity (heart failure) remains a major clinical problem with a poor prognosis and the search for novel treatments remains an important area of research.

Urocortins are proteins that appear to increase blood flow and heart pumping activity. There has been particular interest in the role of Urocortins 2 & 3 (subtypes of Urocortins) in heart failure.

In this study, we will examine the effects and mechanisms of Urocortins 2 & 3 and the Corticotrophin Releasing Hormone Receptor Type 2 (CRH-R2) receptor (through which urocortins act) on forearm blood flow and release of natural blood clot dissolving factors in the forearm circulation of healthy volunteers.

In this study, we will look at the role of the lining of the blood vessel (endothelium) in response to urocortin types 2 and 3. We hypothesise that urocortins 2 & 3 act via the endothelium to cause dilatation of the blood vessels and release of tissue-plasminogen activating factor (blood clot dissolving factor). We also hypothesise that urocortins have a role in maintaining the normal baseline level of blood flow in forearm arteries. In addition to the above, we will also look at the effect of temporarily blocking the effect of urocortins, using a specially designed blocker drug (Astressin 2B).

Utilising the well-established technique of 'forearm venous occlusion plethysmography', we will be able to focus on the local effects of urocortins on arterial blood flow in forearm vessels, without affecting this system in the body as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 - 65 years (inclusive)

Exclusion Criteria:

* Lack of informed consent- Age <18 years > 65 years
* Current involvement in a clinical trial
* Severe or significant co-morbidity including bleeding diathesis, renal or hepatic failure
* Smoker
* History of anaemia
* Recent infective/inflammatory condition
* Recent blood donation (prior 3 months)
* Positive baseline urine test for drugs of abuse (including cannabinoids, benzodiazepines, opiates, cocaine and amphetamines)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-08 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow | 2.30 hours
  Difference between forearm blood flow in response to doses of Ucn2, Ucn3 and Substance P in the presence vs absence of Astressin 2B dose 1 and in the presence vs absence of Astressin 2B dose 2

SECONDARY OUTCOMES:
Net t-PA release | 2.30 hours
  Net t-PA release induced by Ucn2 and Ucn3 in the presence vs absence of Astressin 2B dose 1 and in the presence vs the absence of Astressin 2B dose 2.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Wellcome Trust Clinical Research Facility, Royal Infirmary of Edinburgh, Edinburgh, Mid Lothian, United Kingdom